CLINICAL TRIAL: NCT06082778
Title: Eating Alive: ZOE's Ferment Experiment
Brief Title: ZOE's Ferment Experiment
Acronym: ZHS-FE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zoe Global Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZHS-FE
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Mood; Hunger; Energy
Keywords: Energy; Fermented Foods; Hunger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Increased fermented food intake (Experimental): Participants take part in a n-of-1 design. They are first required to consume their habitual diet, for one week, followed by a period of dietary advice, for two weeks.
  Interventions: Behavioral: Fermented food intake above habitual level

INTERVENTIONS:
Behavioral: Fermented food intake above habitual level — Participants increase their habitual intake of fermented foods by three portions per day, compared to their habitual intake level at baseline.

SUMMARY:
It is not known if an increase in fermented food intake relative to an individuals' habitual diet can lead to improvements in bloating, mood, or hunger levels, or increase energy levels (and reduce fatigue) in the general population. Acceptability of fermented foods across many different types of people and households is also unclear. Therefore, this research aims to investigate the potential effects of increasing fermented food intake on these outcomes, as well as the feasibility of this dietary change.

DETAILED DESCRIPTION:
Background:

Fermented foods (e.g., kombucha, kimchi, sauerkraut) are living foods containing an ecosystem of bacteria and yeasts that use enzymes to process and transform food components. The process of fermentation results in an enhanced nutritional profile of these foods (including probiotics, prebiotics, and additional vitamins) which are associated with health benefits. The majority of people in the Western world consume low amounts of fermented food with live cultures; ~70% report never or rarely consuming fermented foods.

Existing research demonstrates that there are benefits to consuming fermented foods, including improvement of gut microbiome composition as well as reducing inflammation. Furthermore, fermented foods are a unique source of B vitamins that are related to energy levels. Low energy levels are a common but complex problem that affects healthy individuals as well as those with chronic health conditions. Whilst the underlying causes of low energy are unclear, they are a common complaint of many digestive disorders, autoimmune, chronic inflammatory conditions, and metabolic and mood disorders, all of which are associated with disturbance of the gut microbiome. Humans are unable to produce B vitamins and are reliant on diet or gut microbes to produce them. Vitamin B12 levels are ten fold greater in fermented dairy products, and can be found in fermented plant-based foods such as tempeh, making these foods a valuable source of vitamin B12, a nutrient that the human diet is commonly deficient in. Fermented foods may have the potential to improve energy, and mood, by increasing gut diversity and reducing inflammation.

Population:

This research is open to participants who are enrolled in the ZOE Health Study. Participants must be at least 18 years of age and must provide their consent in order to participate.

Design:

The Fermented Foods study will take place in an entirely remote format. This study will take part in two phases. Firstly, the participant will complete a habitual diet phase lasting one week, where the participant reports study outcomes while consuming their habitual diet (including habitual intake level of fermented foods). Secondly, the participant will complete the modification phase lasting two weeks, throughout which they are required to introduce, or increase, their habitual intake of fermented foods by three portions per day (e.g., where a participant normally consumes 1 serving per day, they will now be asked to consume 4 servings per day).

Using the ZOE Health Study app, participants will be asked to:

* Complete questionnaires to assess habitual food intake, dietary habits, health history, sleep, bowel habits and digestive health at the start and end of the study.
* Log levels of hunger, energy, mood and bloating, on a daily basis, throughout the entire study period (baseline and modification phase) using the study app.
* Log their portion intake of fermented foods, on a daily basis, throughout the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* All adults aged 18
* Able to give informed consent
* Are participants of the ZOE Health Study
* Reside in the UK.

Exclusion Criteria: Participants will be excluded if they are:

* Below the age of 18 years.
* Have an histamine intolerance.
* Have a compromised immune system.
* Have been instructed to follow a salt-restricted diet.
* Consume 8 or more portions of fermented foods on a daily basis at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-11-06 (Estimated); Study Completion 2023-11-06 (Estimated)

PRIMARY OUTCOMES:
Daily energy level | 3 weeks
  Participants will self-report their energy level daily using a Visual Analogue Scale ranging from 0 to 10. Higher scores represent better outcomes.

SECONDARY OUTCOMES:
Daily sensation of abdominal bloating | 3 weeks
  Participants will self-report their severity of abdominal bloating daily using a Visual Analogue Scale ranging from 0 to 10. Higher scores represent worse outcomes.
Change in mood | 3 weeks
  Participants will self-report their mood at baseline and wk-3 using a modified version of the Visual Analogue Mood Scale (VAMS) in response to questions about specific mood states (Happy, Sad, Calm, Tense, Energetic, Sleepy). The scale ranges from 0 to 100, with higher scores representing better outcomes for 'Happy', 'Calm' and 'Energetic'; and worse outcomes for 'Sad', 'Tense' and 'Sleepy'.
Daily level of mood | 3 weeks
  Participants will self-report their mood daily, using a Visual Analogue Scale ranging from 0 to 10. Higher scores represent better outcomes.
Change in hunger level | 3 weeks
  Participants will self-report their hunger level at baseline and wk-3, in response to questions about specific hunger symptoms, with answer options following a Likert scale ranging from 'strongly agree' to 'strongly disagree'.
Daily hunger level | 3 weeks
  Participants will self-report their hunger level daily, using a Visual Analogue Scale ranging from 0 to 10. Higher scores represent worse outcomes.

OTHER OUTCOMES:
Change in digestive symptoms | 3 weeks
  Participants will self-report their commonly experienced digestive symptoms and those that they receive treatment for, at both baseline and wk-3.
Change in bowel movements | 3 weeks
  Participants will self-report their average frequency of bowel movements at baseline and wk-3.
Change in stool form | 3 weeks
  Participants will self-report the most common form of their stool form at baseline and wk-3 using the Bristol Stool Form Scale. This scale ranges from 1 to 7, with lower values indicating constipation (1-2), whereas higher values (5-7) may indicate diarrhoea and urgency.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Spector, Pr, Principal Investigator — Zoe Ltd; Will Bulsiewicz, Dr, Principal Investigator — Zoe Ltd
Locations (1):
- ZOE Ltd, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No